CLINICAL TRIAL: NCT00244543
Title: A Single-Center, Double-Masked, Randomized, Placebo-Controlled, Evaluation of the Onset and Duration of Action of R89674 0.25% Ophthalmic Solution in Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis
Brief Title: Evaluation of Efficacy of Ophthalmic Solution in Induced Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-003-13
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Conjunctivitis
Keywords: ocular, allergic conjunctivitis, ophthalmic
MeSH Terms: conditions — Conjunctivitis, Allergic

INTERVENTIONS:
Drug: R89674 (generic name not yet established)

SUMMARY:
The purpose of this study is to establish the efficacy of R89674 0.25% ophthalmic solution compared with placebo in alleviating the signs and symptoms of conjunctival allergen challenge-induced allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

history of ocular allergies and a positive skin test reaction to cat hair, cat dander, grasses, ragweed, and/or trees within the past 24 months; calculated best-corrected visual acuity of 0.6 logMar or better in each eye; positive bilateral conjunctival allergy challenge reaction

-

Exclusion Criteria:

narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium or diagnosis of dry eye; ocular surgical intervention within 3 months; history of refractive surgery within 6 months; known history of retinal detachment, diabetic retinopathy, or progressive retinal disease; presence of active ocular infection positive history of an ocular herpetic infection; preauricular lymphadenopath; manifest signs or symptoms of clinically active allergic conjunctivitis

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110
Dates: Start 2005-10; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Ocular itching and conjunctival redness post challenge

SECONDARY OUTCOMES:
Ciliary and episcieral redness; chemosis; lid swelling; tearing; ocular mucous discharge; and nasal symptoms. All measured postchallenge

CONTACTS AND LOCATIONS:
Overall Officials: Ingerman Avner, MD, Study Director — Johnson & Johnson
Locations (1):
- North Andover, Massachusetts, United States